CLINICAL TRIAL: NCT05437458
Title: Parkinson's Disease: Risk Assessment of Persistent Delirium and Its Management
Acronym: PARADIGM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Other Study IDs: 293560
Record Dates: First submitted 2022-04-04; First posted 2022-06-29 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease; Delirium in Old Age
Keywords: Parkinson's; Delirium; Older
MeSH Terms: conditions — Parkinson Disease; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Persistent delirium: People with Parkinson's who have experienced persistent delirium (delirium lasting for ≥14 days) and will also be invited to interview.
  Interventions: Other: Delirium (exposure)
- Non-persistent delirium: People with Parkinson's who have experienced non-persistent delirium (delirium lasting <14 days).
  Interventions: Other: Delirium (exposure)
- No delirium (Control group): People with Parkinson's who have never experienced delirium
- Carers for Qualitative Interview: Carers of people with Parkinson's who have consented to being interviewed.
  Interventions: Other: Delirium (exposure)

INTERVENTIONS:
Other: Delirium (exposure) — No interventions.
  Groups: Carers for Qualitative Interview; Non-persistent delirium; Persistent delirium

SUMMARY:
Background: delirium describes the change in people's behaviour and thinking when they are unwell. People with delirium may appear confused, have difficulty with organisation and can be different to their usual personality. Older people with Parkinson's are particularly susceptible to persistent delirium, which can last over 14 days. They are more likely to need increased community support and they have a greater risk of death and dementia.

However, there is limited research for people with Parkinson's on how to effectively manage persistent delirium and how to identify those at risk of persistent delirium. Community support may not sufficiently support the care needs of people with Parkinson's, and this is expected to be more detrimental for people also affected by persistent delirium

Study Design: retrospective case note review with qualitative interviews.

Study participants: older people (≥65 years old) with Parkinson's disease, previously affected by either persistent delirium or another form of delirium (e.g. hyperactive, hypoactive, mixed). 207 participants with Parkinson's for quantitative data collection. The qualitative study will include up to 10 participants with Parkinson's from the quantitative part of this study. An additional maximum of 10 more carers for people with Parkinson's may also be interviewed.

Research Aims:

1. To develop and estimate the assessment tool's sensitivity and specificity to predict persistent delirium in older people with Parkinson's in the outpatient setting. Persistent delirium in this study will be initially defined as a delirium lasting ≥14 days. An associated secondary objective will be to develop a scoring system that allocates an increasing number of points to risk factors that have a stronger association for predicting delirium.
2. To evaluate the management strategies used for persistent delirium.
3. To determine what are the community care needs for people recovering from persistent delirium.

DETAILED DESCRIPTION:
Background and Rationale Parkinson's disease is the second most common neurodegenerative condition. Delirium is an acute neuropsychiatric syndrome characterised by an altered level of consciousness, confusion and impaired attention. Usually, delirium is transient if the aetiological factors are corrected or if its effects are minimised by medical treatment. Delirium is potentially preventable in 30-40% of cases, but delirium can result in increased mortality and an increased risk of dementia.

Persistent delirium is when delirium continues to affect patients over weeks to months. However, the exact duration for delirium to be defined as being persistent remains controversial. Previous studies have reported the duration of persistent delirium to be between 7 days to >4 weeks. Persistent delirium in this study will be defined as delirium lasting ≥14 days, which is the average reported by the previous studies. Delirium in older people at the point of hospital discharge is associated with worse outcomes regarding function, cognition, mortality and are more likely to need nursing home placement.

People with Parkinson's could be five times more likely to develop delirium and often delirium in Parkinson's is under-recognised in secondary care.

The use of risk stratification of delirium in people with Parkinson's could highlight the most vulnerable patients so that preventive care can be implemented to minimise their risk of adverse outcomes and complications.

Currently, management strategies for delirium in Parkinson's disease are predominantly based on expert opinion and there is a need for research to determine what are the optimal management strategies for this patient group. Moreover, there are concerns that current community support services do not adequately address the psychosocial issues in older people with advanced Parkinson's disease, which may provide an even greater challenge for patients recovering from persistent delirium.

In summary, older people with Parkinson's are particularly susceptible to delirium, but there is also a paucity of research in this area, which needs to be urgently addressed, to not only prevent the adverse outcomes at an individual level but also the detrimental socio-economic impacts on the wider community.

Participant Recruitment

Eligible potential participants will be invited to the study by their usual medical team during an outpatient Parkinson's clinic at a rural, district general hospital. Eligible potential participants with their permission will be contacted by researchers. Carers of people with Parkinson's will be invited to a qualitative interview. Participants will be recruited consecutively in the order that consent forms were completed till the target sample size has been achieved for the quantitative part of the study. For the qualitative part of the study, recruitment will cease once data saturation has been reached.

Methods

There are 3 main parts to this study:

1. Development and testing of an assessment tool for persistent delirium in people with Parkinson's:

   Participants will be recruited from outpatient clinics for people with Parkinson's this may take up to 8 months. Initially, the potential participant's usual doctor will invite them to take part in the study, before the research team goes through the details of the study with the potential participant.

   Written informed consent will be needed. If the potential participant cannot consent for themselves, then a consultee will be contacted. A consultee is someone that is well known to the potential participant and is willing to advise on whether the potential participant, should take part in the study. In tandem with participant recruitment for at least 14 months, there will be data collection from medical records. Medical records will be reviewed to identify the characteristics and events that have affected people who then go on to develop persistent delirium. Participants' characteristics that will be analysed will be broadly related to their general level of physical fitness, the severity of their Parkinson's disease, visual or hearing difficulties and any conditions affecting their mind, such as dementia.

   Events that the medical notes will be checked for include: the medical care, blood tests and imaging that the participant received, any complications during their hospital stay and the support that they received in the community. Participants will be divided into 3 groups: those with persistent delirium, which is where participants become unwell, which has led to the participant becoming confused or have changes in their behaviour for 14 days or more. Another group with non-persistent delirium, this is when the delirium has lasted less than 14 days and a control group who have not had delirium at all.

   The Chief Investigator will write a summary of each participant but identifiable details will be excluded. These summaries will be reviewed by at least one other medical specialist involved in the care of older people, to double-check that the study findings are as accurate as possible. Potentially, another medical colleague may be required if there is any initial disagreement between specialists. To further confirm the accuracy of the findings, healthcare staff entries in the notes and information collected from relatives/carers can also be used. 8 months will be needed to develop and test the assessment tool.

   This will be done by using statistical methods, such as logistic regression to determine which of these factors are most strongly linked to persistent delirium. A scoring system can be developed, which allocates an increasing number of points to participants with a risk factor that is more strongly linked to persistent delirium. The accuracy of the tool will be determined by its ability to detect people with delirium (sensitivity) and its ability to detect people without delirium (specificity). It is estimated that 207 participants will be required. This is assuming that persistent delirium is present in approximately 20% of patients. The estimate of persistent delirium is based on local audit data.
2. Development of a management plan

   From the information collected in 1), there will be a review of the care that a participant received to identify factors that helped and hindered their recovery from delirium. This information will allow the Chief Investigator to begin to develop a care plan, which can then be tested in future studies. The majority of the data needed will be collected during the development of the assessment tool. The writing up of the study will begin 1 year after the beginning of the study and conclusions will be drawn from these data.

   Data Analysis of Quantitative Data

   The extracted data is expected to be non-parametric. Descriptive statistics will describe participants' demographics and clinical characteristics, using mean, median, standard deviation, interquartile range and percentages.

   The Kruskal-Wallis test will be used to establish if there is a statistically significant difference between two or more groups (e.g. those without delirium, those with non-persistent delirium and those with persistent delirium). Post hoc tests will elucidate which groups differ from each other. Chi-squared tests will compare between-group distributions of proportions. Repeated measures ANOVA or Friedman's will determine changes in repeated measure assessments (e.g. full blood count, urea and electrolytes, c-reactive protein). Hierarchical logistic regression analysis, adjusting for covariates (e.g. demographics, clinical factors, infection), will ascertain the significant risk factors for delirium and provide odds ratios. Multiple comparisons will be corrected using Bonferroni's correction.

   Survival analysis will be utilised to determine the time to the outcomes of interest, such as persistent delirium, mortality and increase in community support. Survival curves will be compared using the log-rank test. It is expected that participants' medical records will have missing data. Missing data will be recorded to determine if there are any missing value patterns, associated with certain outcomes.

   To develop the assessment tool, the "regularised" regression techniques, such as LASSO or Elastic Net will be used. A scoring system will be devised which allocates an increasing number of points to risk factors that have a stronger association for predicting persistent delirium. The sensitivity and specificity of the risk assessment tool will be calculated and these characteristics will be displayed as ROC (Receiver Operator Characteristic) curves. AUC (Area Under the ROC Curve) can summarise the overall accuracy of the test and this can be computed by the trapezoidal rule. Adjusted odds ratios calculated using logistic regression will compare this study's secondary objective: associations between the management of persistent delirium and its outcomes. These findings will be assessed for their suitability for a larger study to be conducted by the Chief Investigator and these data can inform researchers about the sample size requirements for future studies.
3. Interviews

Written informed consent will be sought from people with Parkinson's and their carer when they attend their routine hospital follow-up appointment. A single researcher will then meet with the participant for a one-to-one interview, lasting for about 1 hour. The interview will be conducted at either the participant's own home or another pre-arranged venue. Questions will focus on the participant's experiences of hospital, the care that they received when they returned home and the challenges that they faced in the community. It is expected that up to 20 participants in total are needed for this study, consisting of up to 10 people with Parkinson's and up to 10 carers. The interviews will begin 2 years into the study and participants will be re-consented to ensure that they still agree to the interview.

Data Analysis of Qualitative Data

The qualitative study will be analysed using thematic analysis. Phrases or expressions from the transcripts will be coded to identify interesting features. Open coding will first be used, which allows the early formation of themes and concepts. These early themes will be reviewed by comparing them to other transcripts to refine and develop recurrent themes. From this, the themes will be defined and a thematic coding frame will be produced which will include sub-themes. This process will be data-driven coding and these data will undergo open, axial and selective coding. The constant comparative method will be used to analyse data to develop a grounded theory, to explain some of the participants' behaviours and reactions to persistent delirium. To achieve this, there will simultaneous analysing and coding of data; each new set of data will be compared to previous extracts, new codes and themes will be added as necessary whilst comparing participants' responses, so that the themes are refined. Integration of these findings will begin the development of an explanatory model. Findings will be reported as recommended by COREQ (consolidated criteria for reporting qualitative research) guidance. The Chief Investigator will be the main data coder, with assistance from Co-Investigators.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for People with Parkinson's:

1. Participants must be aged at least 65 years old in 2015.
2. Participants must have a diagnosis of idiopathic Parkinson's disease using Queen's Square Brain Bank criteria (32) diagnosed by a movement disorders expert.
3. Admitted patients must have stayed in hospital >24 hours for at least one hospital admission.
4. Participants must have had previous admissions/attendance to the hospital between 2015-2019.
5. An appropriate consultee must be available and willing to be involved in this study for potential participants without the mental capacity to consent to the extraction of information from their medical records.
6. For the qualitative study, participants must have the mental capacity to consent and must have been affected by persistent delirium. The participant must be able to understand, write and speak English.

Inclusion Criteria for Carers in the Qualitative Study

1. Participants must be aged 18 or over.
2. Participants must have the mental capacity to consent.
3. Participants must have been a primary carer for someone living with Parkinson's, who has had a previous experience of persistent delirium, during 2015-2020.
4. Participants must be able to understand, write and speak English.

Exclusion Criteria:

Exclusion Criteria for People with Parkinson's

1. Aged less than 65 years old in 2015.
2. Diagnosed with drug-induced parkinsonism, vascular parkinsonism, atypical Parkinsonian disorder (e.g. progressive supranuclear palsy, multiple systems atrophy, corticobasal syndrome) or dementia (e.g. dementia with Lewy bodies, vascular dementia, Alzheimer's disease).
3. Potential participants will be excluded from the interview if they cannot communicate verbally or cannot read/write in English.
4. The potential participant's medical records are incomplete and no alternate strategies are appropriate to account for the missing data, without introducing significant study bias or inaccuracy in statistical findings. Criteria for when the medical records will be excluded in the analysis will be:

1. There is uncertainty regarding the identity of the medical records. 2. Documentation for the admission of interest is missing to the extent that researchers are unable to extract the relevant data required for the aims of this study.

5) For the qualitative study, potential participants will be excluded if they do not have the mental capacity to consent.

6) Potential participants without a consultee and also do not have the mental capacity to consent to this study.

7) Potential deceased participants will be excluded if there is previous documentation that the person would not have wanted to participate in research studies.

Exclusion Criteria for Carers in the Qualitative Study

1. The potential participant is aged less than 18 years old.
2. The potential participant does not have the mental capacity to consent to this study.
3. The potential participant is not the primary carer for someone with Parkinson's and has been affected by persistent delirium, during 2015-2020.
4. The potential participant does not understand, write and/or speak English.
5. The potential participant has a severe speech impairment to the extent that the audio recording of the interview is unintelligible.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. People aged 65 years or older in 2015, with a diagnosis of idiopathic Parkinson's, who attend the outpatient clinic at Airedale Hospital and have had a hospital admission of at least 24 hours during 2015-2019.
  2. A carer (aged 18 years and older) for a person with Parkinson's, who has experienced persistent delirium.
Sampling Method: Probability Sample
Enrollment: 217 (Estimated)
Dates: Start 2022-02-06 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and prevalence of delirium in older people with Parkinson's, measured by the DSM-V criteria (Diagnostic and Statistical Manual of Mental Disorders 5th edition). | Time frame: measured when the participant has previously encountered healthcare professionals during 2015-2019.
  DSM-V (Diagnostic and Statistical Manual of Mental Disorders 5th edition) will be used to confirm the diagnosis of delirium.
The duration of delirium will be measured in days. | Time frame: measured when the participant has previously encountered healthcare professionals during 2015-2019.
  Once delirium is confirmed by the DSM-V criteria, then the number of days that participants are affected by delirium will be inferred from medical notes.

CONTACTS AND LOCATIONS:
Overall Officials: William Lee, MB/BS, Principal Investigator — Airedale Hospital
Locations (1):
- Airedale Hospital, Keighley, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
To occur after the PARADIGM has published its study findings.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At after 2025 for at least 5 years.
Access Criteria: By written request to principal investigator.

REFERENCES:
- [Background] AMERICAN PSYCHIATRIC ASSOCIATION 2013. Delirium. Diagnostic and statistical manual of mental disorders. 5th ed. Washington, DC.
- [Background] Billings J, Mijanovich T. Improving the management of care for high-cost Medicaid patients. Health Aff (Millwood). 2007 Nov-Dec;26(6):1643-54. doi: 10.1377/hlthaff.26.6.1643. PMID 17978384
- [Background] BRAUN, V. & CLARKE, V. 2006. Using thematic analysis in psychology. Qualitative research in psychology, 3, 77-101.
- [Background] Cole MG, Ciampi A, Belzile E, Zhong L. Persistent delirium in older hospital patients: a systematic review of frequency and prognosis. Age Ageing. 2009 Jan;38(1):19-26. doi: 10.1093/ageing/afn253. Epub 2008 Nov 18. PMID 19017678
- [Background] Davis DH, Muniz Terrera G, Keage H, Rahkonen T, Oinas M, Matthews FE, Cunningham C, Polvikoski T, Sulkava R, MacLullich AM, Brayne C. Delirium is a strong risk factor for dementia in the oldest-old: a population-based cohort study. Brain. 2012 Sep;135(Pt 9):2809-16. doi: 10.1093/brain/aws190. Epub 2012 Aug 9. PMID 22879644
- [Background] Kakuma R, du Fort GG, Arsenault L, Perrault A, Platt RW, Monette J, Moride Y, Wolfson C. Delirium in older emergency department patients discharged home: effect on survival. J Am Geriatr Soc. 2003 Apr;51(4):443-50. doi: 10.1046/j.1532-5415.2003.51151.x. PMID 12657062
- [Background] Kouli A, Torsney KM, Kuan WL. Parkinson's Disease: Etiology, Neuropathology, and Pathogenesis. In: Stoker TB, Greenland JC, editors. Parkinson's Disease: Pathogenesis and Clinical Aspects [Internet]. Brisbane (AU): Codon Publications; 2018 Dec 21. Chapter 1. Available from http://www.ncbi.nlm.nih.gov/books/NBK536722/ PMID 30702842
- [Background] Lawson RA, McDonald C, Burn DJ. Defining delirium in idiopathic Parkinson's disease: A systematic review. Parkinsonism Relat Disord. 2019 Jul;64:29-39. doi: 10.1016/j.parkreldis.2018.09.025. Epub 2018 Sep 26. PMID 30279060
- [Background] Lubomski M, Rushworth RL, Tisch S. Hospitalisation and comorbidities in Parkinson's disease: a large Australian retrospective study. J Neurol Neurosurg Psychiatry. 2015 Mar;86(3):324-30. doi: 10.1136/jnnp-2014-307822. Epub 2014 May 29. PMID 24876185
- [Background] MEHRA, A., SURENDRAN, I., SURI, V. & GROVER, S. 2014. Missed diagnosis-persistent delirium. Journal of Geriatric Mental Health, 1, 118.
- [Background] Read J, Cable S, Lofqvist C, Iwarsson S, Bartl G, Schrag A. Experiences of health services and unmet care needs of people with late-stage Parkinson's in England: A qualitative study. PLoS One. 2019 Dec 30;14(12):e0226916. doi: 10.1371/journal.pone.0226916. eCollection 2019. PMID 31887175
- [Background] Siddiqi N, House AO, Holmes JD. Occurrence and outcome of delirium in medical in-patients: a systematic literature review. Age Ageing. 2006 Jul;35(4):350-64. doi: 10.1093/ageing/afl005. Epub 2006 Apr 28. PMID 16648149
- [Background] ROSNER, B. 2015. Fundamentals of biostatistics, Cengage learning.
- [Background] TAYLOR, S. J. & BOGDAN, R. 1984. Introduction to qualitative research methods: The search for meanings, Wiley-Interscience.
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Frank M, Sivagnanaratnam A, Bernstein J. Nutritional assessment in elderly care: a MUST! BMJ Qual Improv Rep. 2015 Jan 22;4(1):u204810.w2031. doi: 10.1136/bmjquality.u204810.w2031. eCollection 2015. PMID 26734346
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Kuhn E, Du X, McGrath K, Coveney S, O'Regan N, Richardson S, Teodorczuk A, Allan L, Wilson D, Inouye SK, MacLullich AM, Meagher D, Brayne C, Timmons S, Davis D. Validation of a consensus method for identifying delirium from hospital records. PLoS One. 2014 Nov 4;9(11):e111823. doi: 10.1371/journal.pone.0111823. eCollection 2014. PMID 25369057